CLINICAL TRIAL: NCT05871970
Title: A Phase 2a/b Single Arm Open Label Study to Evaluate the Safety and Efficacy of Intracystic Administration of TARA-002 in Participants Between 6 Months to Less Than 18 Years of Age for the Treatment of Macrocystic and Mixed Cystic Lymphatic Malformations
Brief Title: Safety and Efficacy Study of Intracystic TARA-002 for the Treatment of Lymphatic Malformations in Participants 6 Months to Less Than 18 Years of Age
Acronym: STARBORN-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Protara Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARA-002-201
Record Dates: First submitted 2023-05-11; First posted 2023-05-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Lymphatic Malformation
Keywords: Macrocystic lymphatic malformations; Mixed-cystic lymphatic malformations
MeSH Terms: conditions — Lymphatic Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TARA-002 (Experimental): TARA-002 is a lyophilized biological preparation for injection containing cells of Streptococcus pyogenes (Group A, type 3) Su strain treated with benzylpenicillin.
  Interventions: Biological: TARA-002

INTERVENTIONS:
Biological: TARA-002 — All participants will receive up to 4 intracystic injections spaced approximately 6 weeks apart.

SUMMARY:
This is a Phase 2a/b single arm open label study to evaluate the safety, reactogenicity, and efficacy of intracystic injection of TARA-002 in participants 6 months to less than 18 years of age for the treatment of macrocystic and mixed cystic lymphatic malformations. The Phase 2a safety lead-in, age de-escalation study is designed to establish the safety of TARA-002 in older participants 6 years to less than 18 years before proceeding to younger participants 2 years to less than 6 years, then 6 months to less than 2 years. The Phase 2b is an expansion study in which enrollment of participants will be initiated after safety has been established in each cohort during the Phase 2a safety lead-in study. Each participant will receive up to 4 injections of TARA-002 spaced approximately 6 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 6 months to less than 18 years of age at the time of informed consent/assent form was signed
* Participants whose parent/LAR(s) have voluntarily given written consent and participants who provided assent (if applicable) after the study has been explained to them
* Participants with macrocystic LM or mixed cystic LM (≥ 50% macrocystic disease measured by volume) of the Head/Neck/Mediastinum according to the ISSVA 2018 criteria (ISSVA 2018) measured via LM imaging at Screening to confirm, upon central review, the diagnosis of macrocystic or mixed cystic LM
* Participants who may have had surgical or sclerotherapy treatment for their LM, but not within six months of the consent/assent form being signed

Exclusion Criteria:

* Penicillin allergy
* Vascular tumors or combined vascular malformations
* Microcystic LM or mixed cystic LM with predominant microcystic features
* LMs of the orbit (orbital LM) as target cyst

For more information on eligibility criteria, please contact the sponsor.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with clinical success after one treatment cycle of TARA-002 | 8 weeks after the last injection

SECONDARY OUTCOMES:
Safety: Percentage of participants with solicited local site and systemic reactions | 14 days (2 weeks) after each injection
Safety: Percentage of participants with unsolicited adverse events (AEs) | Through study completion (approximately 32 weeks after last injection)
Safety: Percentage of participants with SAEs, AEs of special interest, AEs leading to premature discontinuation of study intervention, AEs leading to withdrawal from study, AEs with an outcome of death, and MAAEs | Through study completion (approximately 32 weeks after last injection)
Durable Response: Proportion of participants with clinical success after one treatment cycle of TARA-002 assessed at 8 weeks after the last injection and maintained clinical success at 32 weeks after the last injection | 32 weeks after the last injection
Clinical Success by LM Type: Proportion of participants with macrocystic LM or mixed cystic LM with clinical success after one treatment cycle of TARA-002 | 8 weeks after the last injection
Investigator Assessment: Proportion of participants who demonstrate clinical improvement, as assessed by the Investigator, after one treatment cycle of TARA-002 compared to baseline | 8 weeks after last injection and 32 weeks after last injection
Quality of Life: Change in Quality-of-Life assessment based on Pediatric Quality of Life Inventory (PedsQL) and Visual Analog Scale (VAS) for Pain after one treatment cycle of TARA-002 | 8 weeks after last injection and 32 weeks after last injection

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Operations Officer, Study Director — Protara Therapeutics
Locations (10):
- United States (10):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital/UAMS, Little Rock, Arkansas
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center: Children's Research Institute, Washington D.C., District of Columbia
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia: Comprehensive Vascular Anomalies Program, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Hospital of the King's Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No